CLINICAL TRIAL: NCT04915573
Title: Antimicrobial Resistance Among Sputum Pathogens in Post Hepatitis Cirrhotic Patients
Brief Title: Antimicrobial Resistance in Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer, Mansoura University
Other Study IDs: 34647/4/21
Record Dates: First submitted 2021-05-29; First posted 2021-06-07 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — sputum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Cirrhosis: Patient with clinical evidence of liver disease, portal hypertension, ultrasound or computed tomography results, laboratory data will be used to confirm liver disease
  Interventions: Diagnostic Test: Specimen

INTERVENTIONS:
Diagnostic Test: Specimen — Sputum will be collected in clean disposable containers

SUMMARY:
Cirrhotic patients are more vulnerable to bacterial infection, and infection is one of the most common causes of acute liver disease decompensation.

DETAILED DESCRIPTION:
Cirrhotic patients are more vulnerable to bacterial infection which is a common cause of acute liver disease decompensation. The aim of this study will characterize the antimicrobial resistance and distribution of bacteria isolated from chronic hepatic patients with pulmonary infections, as well as to evaluate the antimicrobial susceptibility of bacteria isolated from sputum.

ELIGIBILITY:
Inclusion Criteria:

1. Adults' older than 18 years with clinical evidence of liver disease

Exclusion Criteria:

1. Pregnancy
2. Intensive care unite stay of more than 24 hours
3. Malignancy
4. Organ transplantation
5. Acquired immune deficiency syndrome

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Isolate Identification | One day
  Distribution of bacterial isolates from sputum of cirrhotic patients expressed by frequency of each isolate
Antimicrobial resistance | One day
  Antimicrobial susceptibility testing to antibiotics determined by kirby-bauer disk diffusion

CONTACTS AND LOCATIONS:
Overall Officials: Noha Mansour, Ph.D, Study Director — Mansoura University
Locations (1):
- Tanta University Hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided